CLINICAL TRIAL: NCT05125328
Title: To Explore the Optimal Dose of Remifentanil for Skull Pin Fixation in Intracranial Surgery.
Brief Title: ANI and Remifentanil in Skull Pin Fixation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20210156
Record Dates: First submitted 2021-10-11; First posted 2021-11-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pain, Procedural
Keywords: remifentanil; pain; analgesia nociception index
MeSH Terms: conditions — Pain, Procedural; Pain | interventions — Remifentanil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- neurosurgery with fixation (Experimental)
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Remifentanil — First start with remifentanil 6.0 ng/ml, and use the up and down method as adjust 0.5 ng/ml of concentration of remifentanil each time. An ANI lower than 30 and hyperdynamics (the increased heart rate and mean blood pressure up 20% of baseline or heart rate>100bpm and arterial blood pressure>180/100mmHg) indicates insufficient analgesia, therefore increase it by 0.5 ng/ml; an ANI higher than 30 and stable hemodynamics (the changes of HR and MBP within 20% of baseline or HR<50bpm and ABP<90/50mmHg) indicates that analgesia is acceptable, and the next patient will decrease it by 0.5 ng/ml during skull pin fixation.

SUMMARY:
Forty patients were enrolled, and all patients used total intravenous anesthesia (remifentanil-propofol based total intravenous analgesia) as anesthesia induction and maintenance. According to the preliminary data of this department, patients who underwent intracranial surgery for skull pin fixation used remifentanil 5.0-6.0 ng/ml, while the hemodynamics is relatively stable. Therefore, when this plan is implemented, the patient needs to be under the same depth of anesthesia (monitored by electroencephalography, maintaining a value of 40-60), first start with remifentanil 6.0 ng/ml, and use the up and down method as adjust 0.5 ng/ml of concentration of remifentanil each time. An Analgesia Nociception Index(ANI) lower than 30 and hyperdynamics (the increased heart rate(HR) and mean blood pressure(MBP) up 20% of baseline or HR>100bpm and arterial blood pressure(ABP)>180/100mmHg) indicates insufficient analgesia, therefore increase it by 0.5 ng/ml; an ANI higher than 30 and stable hemodynamics (the changes of HR and MBP within 20% of baseline or HR<50bpm and ABP<90/50mmHg) indicates that analgesia is acceptable, and the next patient will decrease it by 0.5 ng/ml during skull pin fixation.

Data collection: Heart Rate, Measure blood pressure, Analgesia Nociception Index, Bispectral index, concentrations of propofol and remifentanil before 2 mins, during, 5, and 15 mins of skull pin fixation were recorded and analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Must be at least 20 years old and less than 80 years old
2. With anesthesia risk grade below grade three (including grade three) (ASA I~III)
3. Patients who are expected to undergo intracranial surgery for skull pin fixation

Exclusion Criteria:

1. Those with anesthesia risk classification ASA class IV or higher
2. Those who are allergic to opioid analgesics or propofol drugs
3. Emergency patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
50% effect concentration of remifentanil | peri-fixation period
  50% effect concentration of remifentanil will be recorded at 2 mins before fixation, during fixation, 5mins after fixation, and 15 mins after fixation.
90% effect concentration of remifentanil | peri-fixation period
  90% effect concentration of remifentanil will be recorded at 2 mins before fixation, during fixation, 5mins after fixation, and 15 mins after fixation.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan